CLINICAL TRIAL: NCT01082237
Title: Biomarkers for Outcomes In Late-life Depression
Brief Title: Biomarkers for Outcomes In Late-life Depression (BOLD)
Acronym: BOLD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ian A. Cook, M.D., Ian A. Cook, M.D., National Institute of Mental Health (NIMH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1RC1MH088438 (NIH); 1RC1MH088438 (NIH)
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; EEG; SSRI
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- escitalopram (Active Comparator): All subjects will receive escitalopram (ESC), brand name Lexapro (Forest Laboratories, Inc., New York) throughout the study. Dosing will start at 5 mg/d, be titrated to 10 mg after 4 days, and continue at 10 mg/d thereafter; an additional dose titration to 20 mg will be pursued at week 8 for those not significantly better (<50% improvement on IDS-30 at week 8 visit) and as tolerated.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Start at 5mg per day, after four days increase to 10mg per day for the duration of the study. 20 mg will be administered at week 8 if not significantly better.
  Other Names: Lexapro

SUMMARY:
Major depressive disorder (MDD) is a common psychiatric illness with high cost to society and individual patients. One reason for the high cost is that most patients endure lengthy and ultimately unsuccessful empiric antidepressant trials before a successful medication is identified by trial-and-error. Care would be improved if a biomarker could determine, early in the course of treatment, whether a particular antidepressant would likely lead to response, remission, or treatment failure. Physicians could rapidly change treatments to an antidepressant which the biomarker indicated would be likely to help the patient. We have identified quantitative electroencephalographic (QEEG) changes that emerge early in the course of treatment with selective serotonin reuptake inhibitors (SSRIs) that appear to predict later response and remission in a general adult patient population. Demographic trends in the United States suggest that improved care for MDD will be essential for a growing number of elderly with late-life depression. While the consequences of prolonged trial-and-error periods to find a successful treatment are particularly inauspicious for elders with late-life depression, this patient group has not been included in the past studies which demonstrated the use of this biomarker approach in a general adult population. We propose a 12-week treatment trial to evaluate a practical biomarker for predicting outcome based on data from the first week of antidepressant treatment, with a focus only on depression in late life (age ≥65).

There are three study Hypothesis:

H1) ATR prediction of treatment outcome in older subjects will show >70% accuracy.

H2) The predictive accuracy of the model will be enhanced by including clinical, socio-demographic, and genetic predictors.

H3) The accuracy of ATR prediction will not show a significant dependence on subject gender.

ELIGIBILITY:
Inclusion Criteria:

* 62 years of age or older
* Meet the DSM-IV diagnosis of MDD based on Sheehan's Mini-International Neuropsychiatric Interview (MINI), with a score of > 28 on the 30-item Inventory of Depressive Symptomatology - Self Rated version (IDS-SR30)

Exclusion Criteria:

* Subjects will have no unstable medical illness that would prevent completion of participation in the trial, determined as needed from physical examination, ECG, laboratory safety tests, as well as a review of systems
* mentally or legally incapacitated, unable to give informed consent
* meets DSM-IV criteria for anorexia nervosa, bulimia nervosa, obsessive-compulsive disorder, any cognitive disorder, bipolar disorder, psychotic disorder, or major depression with psychotic features
* MMSE (Folstein et al., 1975) score ≤ 24
* evidence of drug dependency or substance abuse within the preceding nine months
* stable and in remission on current psychotropic medication(s)
* any ECT within the past six months
* failure to tolerate ESC or treatment failure with an adequate trial of ESC in the current episode
* ESC would be contraindicated (e.g., hyponatremia with a prior SSRI)
* treatment with fluoxetine or an MAOI within the past four weeks
* any medical illness severe enough to significantly affect brain function or to interfere with interpretation of study results
* history of seizures, brain surgery, skull fracture, significant head trauma, or abnormal EEG
* psychiatric hospitalization indicated (e.g., imminent danger to self or others)
* initial QEEG recording is contaminated with artifact so that determination of the biomarker is precluded
* use of medications known to affect brain function (e.g., antidepressants, anticonvulsants/mood stabilizers, anticholinergics, antipsychotics, benzodiazepines - same list as in BRITE-MD)

Min Age: 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Score on Hamilton Depression Rating Scale (HAM-D) | Measured nine times over 8 weeks

SECONDARY OUTCOMES:
Score on Inventory of Depressive Symptomatology-Clinician Rated (IDS-C30) | Measured nine times over 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Cook, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States

REFERENCES:
- See also: Depression — http://www.nlm.nih.gov/medlineplus/depression.html
- See also: Escitalopram — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet